CLINICAL TRIAL: NCT03459378
Title: Retrospective Analysis of Outcome After Implantation of a Transjugular Intrahepatic Portosystemic Shunt (TIPS)
Brief Title: Outcome After TIPS
Status: Completed | Type: Observational
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Other Study IDs: Retro-TIPS
Record Dates: First submitted 2018-02-26; First posted 2018-03-08 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Hypertension, Portal; Liver Cirrhosis; Variceal Hemorrhage; Ascites Hepatic
MeSH Terms: conditions — Hypertension, Portal; Liver Cirrhosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention - retrospective analyses — retrospective data examination, there are no study related interventions

SUMMARY:
This clinical trial is a retrospective single-centre study. Research data will be acquired via patient histories stored in the hospital data system. Data of patients who received a Transjugular Intrahepatic Portosystemic Shunt (TIPS) at the University Hospital Graz between 1.1.2004 and 31.12.2017 will be included into the study. The aim is to investigate the outcome (transplantation free survival, time to (re)occurrence of ascites, occurrence of hepatic encephalopathy) of patients with portal hypertension after TIPS.

DETAILED DESCRIPTION:
The implantation of a Transjugular Intrahepatic Portosystemic Shunt (TIPS) is a valuable measure to reduce portal hypertension and prevent portal hypertension-related complications. It can be used as a symptomatic treatment in patients with chronic portal hypertension as well as for the treatment of active variceal bleedings or large gastrointestinal varices that go along with threatening bleeding danger.

However, this invasive procedure carries a high risk for complications. 30-days mortality after TIPS implantation amounts between 4% and 45%.

A common complication is the (initial) manifestation or deterioration of hepatic encephalopathy, which occurs in 33-46 % after TIPS implantation.

Other complications that are directly related to the intervention are bleeding, infections and stent migration.

Aim of this retrospective single centre study is to investigate the long-term outcome after TIPS implantation with regard to transplantation free survival and time to (re-) occurrence of portal hypertension-related complications, especially ascites and hepatic encephalopathy.

Intervention-related complications as well as long-term effects should be evaluated to facilitate the decision for or against TIPS.

ELIGIBILITY:
Inclusion Criteria:

* every person at the age of 18-90 years who received a Transjugular Intrahepatic Portosystemic Shunt at the University Hospital of Graz/Austria between 1.1.2004 and 31.12.2017

Exclusion Criteria:

* age under 18

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at the age of 18-90 years who received a Transjugular Intrahepatic Portosystemic Shunt at the University Hospital of Graz/Austria between 1.1.2004 and 31.12.2017
Sampling Method: Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2020-05-14 (Actual)

PRIMARY OUTCOMES:
transplantation free survival | from date of TIPS until the event, up to 4 years
  Survival without liver Transplantation in days

SECONDARY OUTCOMES:
occurrence of hepatic encephalopathy | from date of TIPS until the event, up to 4 years
  time to occurrence of the first episode of hepatic encephalopathy in days
occurrence of ascites | from date of TIPS until the event, up to 4 years
  time to (re)occurrence of ascites in days

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Furschuss L, Rainer F, Effenberger M, Niederreiter M, Portugaller RH, Horvath A, Fickert P, Stadlbauer V. A novel score predicts mortality after transjugular intrahepatic portosystemic shunt: MOTS - Modified TIPS Score. Liver Int. 2022 Aug;42(8):1849-1860. doi: 10.1111/liv.15236. Epub 2022 Apr 1. PMID 35261130